CLINICAL TRIAL: NCT07316400
Title: Protocol for a Randomized, Single-Blind, Controlled Clinical Trial Evaluating the Effect of Peptide Polysaccharide Supplementation on Serum Malondialdehyde, Interleukin-6, and Cotinine Levels
Brief Title: PsP Ganoderma Lucidum Supplementation and Biomarker Changes in Smokers
Acronym: PSPGL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brawijaya (Other)
Responsible Party: Principal Investigator, Titin Andri Wihastuti, Principal Investigator (Professor), University of Brawijaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12757/UN10.F17.10.4/TU/2024; 01884.4/UN10.A0501/B/KS/2025 (Other Grant/Funding Number: University of Brawijaya)
Record Dates: First submitted 2025-12-03; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Oxidative Stress; Inflammation; Cigarette Smoking
Keywords: Peptide Polysaccharide (PsP); Ganoderma lucidum; β-Glucan; Oxidative Stress; Inflammation; Smokers
MeSH Terms: conditions — Inflammation; Cigarette Smoking

STUDY DESIGN:
Intervention Model Description: A two-arm parallel design in which adult smokers are randomly assigned to either a control group (smokers without supplementation) or an intervention group (smokers receiving peptide polysaccharide supplementation). Both groups are followed concurrently throughout the study period.
Who Masked: Participant
Masking Description: Participants were blinded to group allocation, with PsP and placebo capsules identical in appearance and packaging. Investigators conducting laboratory analyses were also blinded to group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smoker Control Group (No Supplementation) (No Intervention): Participants in this arm are smokers who do not receive any investigational product. They continue with their usual daily habits without additional supplements or treatments. This group serves as the control for evaluating the effects of PsP Ganoderma lucidum.
- Smokers Receiving PsP Ganoderma lucidum Supplementation (Experimental): Participants in this arm are smokers who receive PsP Ganoderma lucidum as the investigational intervention. They follow the assigned PsP supplementation regimen for the full study duration to assess its effects compared with the control group.
  Interventions: Dietary Supplement: PsP

INTERVENTIONS:
Dietary Supplement: PsP — PsP is a freeze dried Ganoderma lucidum Polysaccharide Peptide extract from mycelium cell wall. Each capsule contains 250 mg of Polysaccharide Peptide, which it equal to 180 mg β-1,3/1,6-D-Glucan.
  Arms: Smokers Receiving PsP Ganoderma lucidum Supplementation

SUMMARY:
The goal of this randomized controlled clinical trial is to evaluate whether polysaccharide peptide (PsP) supplementation from Ganoderma lucidum can modulate biomarkers of oxidative stress, inflammation, nicotine exposure, and stress response in adults exposed to cigarette smoke. The study is conducted in adults aged 20-50 years with active or passive exposure to cigarette smoke.

The main questions it aims to answer are:

* Does PsP supplementation change serum malondialdehyde (MDA) and superoxide dismutase (SOD) levels over 8 weeks?
* Does PsP supplementation affect serum interleukin-6 (IL-6), nitric oxide (NO), cotinine, nicotinic acetylcholine receptor (nAChR), and cortisol levels?

Researchers will compare participants receiving PsP supplementation with those receiving a placebo to evaluate differences in changes in the specified biomarkers.

Participants will:

* Be randomly assigned to receive PsP capsules (500 mg/day) or placebo for 8 weeks
* Provide fasting blood samples at baseline and at the end of the intervention
* Maintain usual lifestyle habits while avoiding antioxidant supplements during the study period

DETAILED DESCRIPTION:
Cigarette smoke exposure is associated with increased oxidative stress and inflammatory responses, largely mediated by excessive production of reactive oxygen species. These processes contribute to elevated levels of lipid peroxidation products and proinflammatory cytokines, as well as measurable biomarkers of nicotine exposure and stress-related physiological responses. Individuals with active or passive exposure to cigarette smoke may therefore experience sustained biochemical alterations linked to oxidative and inflammatory burden.

Polysaccharide peptide (PsP) derived from Ganoderma lucidum is composed primarily of β-(1,3)/(1,6)-D-glucans and peptide fractions that have demonstrated antioxidant and immunomodulatory activity in experimental and preclinical studies. Despite growing interest in PsP as a functional nutritional supplement, clinical evidence evaluating its effects on oxidative stress and inflammation in smoke-exposed human populations remains limited.

This randomized, single-blind, placebo-controlled clinical trial is designed to assess the effects of PsP supplementation on selected serum biomarkers related to oxidative stress, inflammation, nicotine exposure, and stress response. Eligible participants are adults aged 20-50 years with documented active or passive exposure to cigarette smoke. Participants are randomly assigned in a 1:1 ratio to receive either PsP supplementation or a visually identical placebo for a period of 8 weeks.

Participants assigned to the intervention group receive PsP capsules at a total daily dose of 500 mg, administered as one 250 mg capsule twice daily. Each capsule contains standardized amounts of total polysaccharides, including β-glucans, and peptide fractions. The control group receives placebo capsules containing inert excipients with no known biological activity. All study products meet applicable pharmacopeial standards for quality and safety. Adherence to the intervention is monitored through capsule counts and participant-maintained compliance logs.

Fasting blood samples are collected at baseline and at the end of the intervention period. Serum is separated and stored under controlled conditions until analysis. Laboratory assessments are planned using validated analytical methods to quantify biomarkers of oxidative stress, antioxidant activity, inflammation, nicotine exposure, receptor-related parameters, and stress-related hormones.

The primary outcome measures include changes in serum malondialdehyde (MDA) and superoxide dismutase (SOD) concentrations from baseline to week 8. Secondary outcome measures include changes in serum interleukin-6 (IL-6), nitric oxide (NO), cotinine, nicotinic acetylcholine receptor (nAChR) levels, and cortisol concentrations over the same period.

The planned statistical analysis includes descriptive summaries of baseline characteristics and inferential analyses to compare changes in outcome measures between study groups and within groups over time. Appropriate statistical methods are prespecified to account for baseline variability. All analyses are conducted using two-tailed tests with a prespecified level of statistical significance.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults aged 18 to 60 years.
2. Has smoked regularly for at least the past 12 months.
3. Able and willing to provide written informed consent.
4. Agrees to maintain usual smoking habits during the study period.
5. Able to comply with study procedures and visits.

Exclusion Criteria:

1. Current use of antioxidant supplements, vitamins, herbal supplements, or mushroom- derived products within the last 4 weeks.
2. Diagnosis of chronic inflammatory disease, autoimmune disease, diabetes mellitus, cardiovascular disease, chronic kidney disease, chronic liver disease, or cancer.
3. Acute illness, infection, or fever within the last 14 days.
4. Regular use of anti-inflammatory drugs (NSAIDs, corticosteroids) within the last 4 weeks.
5. Participation in another clinical study within the past 30 days.
6. Pregnant or breastfeeding.
7. Known allergy to Ganoderma lucidum or mushroom-derived compounds.
8. Alcohol dependence or substance abuse other than tobacco.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-10-26 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Serum Malondialdehyde (MDA) Levels | Baseline to 8 weeks
  Serum MDA concentration (nmol/mL) will be measured to assess oxidative stress status in participants receiving PsP compared with the control group
Change in Serum Superoxide Dismutase (SOD) Levels | Baseline to 8 weeks
  Serum SOD concentration (U/mL) will be measured to assess oxidative stress status in participants receiving PsP compared with the control group

SECONDARY OUTCOMES:
Change in Serum Interleukin-6 (IL-6) Levels | Baseline to 8 weeks
  Serum IL-6 concentration (pg/mL) will be measured to evaluate the inflammatory response following PsP supplementation compared with control
Change in Serum Nitric Oxide (NO) Levels | Baseline to 8 weeks
  Serum NO concentration (µmol/L) will be measured to evaluate inflammatory response following PsP supplementation compared with control
Change in Serum Cotinine Levels | Baseline to 8 weeks
  Serum cotinine concentration (ng/mL) will be measured as an objective biomarker of tobacco exposure to assess changes during the study period
Change in Serum Nicotinic acetylcholine receptors (nAChRs) Levels | Baseline to 8 weeks
  Serum nAChRs concentration (ng/mL) will be measured as an objective biomarker of tobacco exposure to assess changes during the study period
Change in Serum Cortisol Levels | Baseline to 8 weeks
  Serum Cortisol concentration will be measured as an objective biomarker of tobacco exposure to assess changes during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Titin A Wihastuti, Professor, Principal Investigator — Brawijaya University
Locations (1):
- University of Brawijaya, Malang, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study does not include a data-sharing plan in the ethics approval or informed consent. Data contain sensitive biomarker and smoking-related information that may pose a re-identification risk for participants. Therefore, IPD will not be made publicly available.

REFERENCES:
- [Background] Kumboyono K, Chomsy IN, Hakim AK, Sujuti H, Hariyanti T, Srihardyastutie A, Wihastuti TA. Detection of Vascular Inflammation and Oxidative Stress by Cotinine in Smokers: Measured Through Interleukin-6 and Superoxide Dismutase. Int J Gen Med. 2022 Sep 16;15:7319-7328. doi: 10.2147/IJGM.S367125. eCollection 2022. PMID 36147199
- [Background] Kumboyono K, Nurwidyaningtyas W, Chomsy IN, Wihastuti TA. Early Detection of Negative Smoking Impacts: Vascular Adaptation Deviation Based on Quantification of Circulated Endothelial Activation Markers. Vasc Health Risk Manag. 2021 Mar 23;17:103-109. doi: 10.2147/VHRM.S296293. eCollection 2021. PMID 33790567
- [Background] Wihastuti TA, Heriansyah T. The inhibitory effects of polysaccharide peptides (PsP) of Ganoderma lucidum against atherosclerosis in rats with dyslipidemia. Heart Int. 2017 Apr 12;12(1):e1-e7. doi: 10.5301/heartint.5000234. eCollection 2017 Jan-Dec. PMID 29114382
- See also: Product information for PsP (Peptide Polysaccharide) Ganoderma lucidum supplement, including composition, manufacturing details, and general product background provided by the manufacturer. — http://www.slhlabs.com/psp/?o=default